CLINICAL TRIAL: NCT04947449
Title: Laser Therapy on Burned Skin
Brief Title: Potential Benefits of Laser Treatment on Skin Blood Flow and Sweating in Burn Survivors
Status: Terminated | Type: Observational
Why Stopped: Recruitment and retention challenges, coupled with our focus changing to a different direction.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Craig Crandall, Professor of Medicine, University of Texas Southwestern Medical Center
Other Study IDs: STU-2021-0241
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Burn Injury
Keywords: laser treatment; laser therapy; skin blood flow; sweating
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: fractional CO2 laser — Standard of care laser treatment of burn-related injuries will be performed. This protocol assesses the effects of those treatments on skin blood flow and sweating responses.

SUMMARY:
The purpose of this study is to examine effects of laser therapy on blood flow and sweating responses in burn-injured skin.

DETAILED DESCRIPTION:
This is a longitudinal study in which the effects of laser therapy on cutaneous vascular responses and sweating of the treated areas are assessed. Specifically, burn survivors who will undergo standard of care laser therapy to treat burn-related scars will perform whole-body heating and local heating procedures prior to the initiation of laser therapy, at an intermediate point during the laser therapy regimen, and upon conclusion of the laser therapy regimen.

For this pilot investigation a placebo will not be incorporated.

Primary outcome variables will be skin blood flow and sweating responses from skin treated with laser therapy and adjacent untreated/uninjured skin.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Experience a severe burn injury that warrant laser therapy.
* Free of any significant underlying medical problems based upon a detailed medical history and physical exam

Exclusion Criteria:

* Known heart disease
* Other chronic medical conditions requiring regular medical therapy including cancer, diabetes, uncontrolled hypertension, and uncontrolled hypercholesterolemia.
* Abnormality detected on routine screening suggestive of cardiac ischemia or previously undetected cardiac disease or resting left bundle branch block on screening electrocardiogram.
* Subject with a body mass index >35 kg/m2
* Pregnant or planning to become pregnant within the subsequent 6 months.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy individuals who undergo laser treatment for burn injuries
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Skin blood flow | Upwards to 6 months after the final laser treatment
  Primary outcome variables will be skin blood flow and sweating responses from skin treated with laser therapy and adjacent untreated/uninjured skin.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States